CLINICAL TRIAL: NCT00002993
Title: Evaluation of Mitomycin, Doxorubicin and Cisplatin in the Treatment of Recurrent or Advanced Uterine Sarcomas
Brief Title: Combination Chemotherapy in Treating Patients With Recurrent or Advanced Cancer of the Uterus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000065540; GOG-87I
Record Dates: First submitted 1999-11-01; First posted 2004-09-03 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2006-05

CONDITIONS: Sarcoma
Keywords: stage III uterine sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Cisplatin; Doxorubicin; Mitomycin

INTERVENTIONS:
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: mitomycin C

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy with mitomycin, doxorubicin, and cisplatin in treating patients with recurrent or advanced cancer of the uterus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the antitumor activity of the combination of mitomycin, doxorubicin, and cisplatin (MAP) in patients with recurrent or advanced uterine sarcomas. II. Determine the nature and degree of toxicity of MAP chemotherapy in this cohort of patients.

OUTLINE: Patients receive IV doxorubicin, mitomycin, and cisplatin over 3 hours once every 3 weeks, for a minimum of 1 course. Patients who have complete response, partial response, or stable disease will continue for at least 3 courses. If side effects are not severe, patients may remain on the study regimen at the investigator's discretion for a maximum of 6 courses. All patients are followed until death.

PROJECTED ACCRUAL: The first stage of accrual is anticipated to accrue 20 evaluable patients in approximately 12 months. If indicated, a second stage will accrue approximately 10 evaluable patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced, persistent, or recurrent uterine sarcoma Documented disease progression after local therapy Measurable disease consisting of abdominal, pelvic, chest, or other masses that can be defined in at least two dimensions by palpation, x-ray, computed tomography or ultrasound

PATIENT CHARACTERISTICS: Age: No age specified Performance status: Karnofsky 50%-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT no greater than 3 times normal Alkaline phosphatase no greater than 3 times normal Renal: Creatinine no greater than 1.5 times normal Cardiovascular: Ejection fraction within institutional normal limits Pulmonary: Not specified Other: No active infection No concurrent second malignancy other than nonmelanoma skin cancer Must be disease free of any prior malignancy for at least 5 years and not received any treatments with chemotherapy or radiation therapy for that malignancy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 6 weeks since radiotherapy Recovered from effects of radiotherapy Surgery: Recovered from effects of surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-08; Primary Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H. Edmonson, MD, Study Chair — Mayo Clinic
Locations (54):
- United States (54):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington

REFERENCES:
- [Result] Edmonson JH, Blessing JA, Cosin JA, Miller DS, Cohn DE, Rotmensch J. Phase II study of mitomycin, doxorubicin, and cisplatin in the treatment of advanced uterine leiomyosarcoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2002 Jun;85(3):507-10. doi: 10.1006/gyno.2002.6661. PMID 12051882